CLINICAL TRIAL: NCT00032474
Title: Ginkgo Biloba Extract and the Insulin Resistance Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000832-01 (NIH)
Record Dates: First submitted 2002-03-21; First posted 2002-03-22 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Ginkgo biloba; type 2 diabetes; platelet function; antioxidant
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ginkgo biloba extract

INTERVENTIONS:
Drug: Ginkgo biloba extract

SUMMARY:
The purpose of this study is to examine whether the ingestion of the herbal dietary supplement Ginkgo biloba extract has any effect on the efficacy of three classes of diabetic medications - (Glucotrol, Glucophage and Actose). Additionally, the study will examine the effect of Ginkgo biloba extract on pancreatic insulin production in non-diabetic subjects between the ages of 20 and 75 years old.

DETAILED DESCRIPTION:
Herbal remedy is popular among those with chronic diseases, who may already be taking several prescription medications, thereby increasing the risk of drug-herb interactions. Ginkgo biloba extract is a popular dietary supplement that is ingested by the general population to enhance mental focus and by the elderly to delay onset of age-acquired loss of cognitive function. In subjects with non-insulin dependent diabetes (NIDDM), ingestion of Ginkgo biloba may decrease efficacy of the hypoglycemic agents and increase whole body insulin resistance. Because aging is a significant risk factor for the development of NIDDM as a result of a progressive decline in pancreatic function, and because the elderly chronically take multiple prescription medications, the increased use of Ginkgo biloba in this population may increase drug-herb interactions. Therefore, we shall examine the effect of Ginkgo biloba on the pancreatic function in the elderly to determine whether it may produce pancreatic dysfunction and a potential for the development of insulinopenia. The results of this study should provide valuable information for designing new therapeutic strategies for the treatment of diseases in the insulin resistance syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus and taking oral diabetes medications - Glucotrol, Glucophage and Actose or Avandia
* Must be able to swallow
* Healthy individuals without diabetes aged 20 to 80 years of age

Exclusion Criteria:

* Type 1 diabetes mellitus
* Type 2 diabetes mellitus taking insulin injections
* Regular use of anti-inflammatory drugs
* Chronic anemia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2001-12; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: George B. Kudolo, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Sciences Center, San Antonio, Texas, United States

REFERENCES:
- [Background] Kudolo GB. The effect of 3-month ingestion of Ginkgo biloba extract on pancreatic beta-cell function in response to glucose loading in normal glucose tolerant individuals. J Clin Pharmacol. 2000 Jun;40(6):647-54. PMID 10868316
- [Background] Kudolo GB. The effect of 3-month ingestion of Ginkgo biloba extract (EGb 761) on pancreatic beta-cell function in response to glucose loading in individuals with non-insulin-dependent diabetes mellitus. J Clin Pharmacol. 2001 Jun;41(6):600-11. doi: 10.1177/00912700122010483. PMID 11402628
- [Background] Kudolo GB. Ingestion of Ginkgo biloba extract accelerates pancreatic function in normal and type II diabetic subjects. Clinical Chemistry 2000; 46 (Suppl) Abstract no. 434.
- [Background] Kudolo GB. Ginkgo biloba increases glucose-stimulated insulin production in diabetic subjects with pancreatic exhaustion. Alternative Therapies in Health and Medicine. 2001; 7:S19.
- [Background] Kudolo GB. Ingestion of Ginkgo biloba extract significantly inhibits collagen-induced platelet aggregation and thromboxane A2 synthesis. Alternative Therapies in Health and Medicine 2001; 7:105.
- [Background] George B. Kudolo, Janet Blodgett. In vitro effects of Ginkgo biloba extract on collagen-induced aggregation and thromboxane B2 synthesis in platelets from type 2 diabetic subjects. International Scientific Conference on Complementary, Alternative & Integrative Medicine Research, April 12-14, 2002. (Journal Of Herbal Pharmacotherapy 3: 5. 2003)
- [Background] George B. Kudolo, Janet Blodgett. Effect of Ginkgo biloba ingestion on arachidonic acid metabolism in the platelets of type 2 diabetic subjects. International Scientific Conference on Complementary, Alternative & Integrative Medicine Research, April 12-14, 2002. (Journal Of Herbal Pharmacotherapy 3: 5. 2003)
- [Background] Wen Wang, Jessica Barrientos, Ryan Elrod, Ken Cusi, Janet Blodgett, George B. Kudolo. Effect of Ginkgo biloba extract on platelet aggregation, thromboxane B2 production and leg blood flow in healthy subjects. First International Conference on Whole Person Healing Conference. Washington, DC, March 28-30, 2003.
- [Background] Kudolo GB, Wang W, Barrientos J, Elrod R, Blodgett J. The ingestion of Ginkgo biloba extract (EGb 761) inhibits arachidonic acid-mediated platelet aggregation and thromboxane B2 production in healthy volunteers. J Herb Pharmacother. 2004;4(4):13-26. PMID 15927922
- [Background] Kudolo GB, Dorsey S, Blodgett J. Effect of the ingestion of Ginkgo biloba extract on platelet aggregation and urinary prostanoid excretion in healthy and Type 2 diabetic subjects. Thromb Res. 2002 Nov 1;108(2-3):151-60. doi: 10.1016/s0049-3848(02)00394-8. PMID 12590952
- [Background] Kudolo GB, Wang W, Dorsey S, Blodgett J. Oral ingestion of Ginkgo biloba extract reduces thiobarbituric acid reacting (TBAR) substances in washed platelets of healthy subjects. J Herb Pharmacother. 2003;3(4):1-15. PMID 15277117